CLINICAL TRIAL: NCT05440409
Title: CAR-Multicenter Analysis (CAR-MA): Retrospective Study to Characterize CAR T-cell Outcomes and Related Toxicities in Children and Young Adults With B-ALL
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000651; 000651-C
Record Dates: First submitted 2022-06-29; First posted 2022-06-30 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06-24

CONDITIONS: Leukemia, Acute Lymphoblastic; Lymphoblastic Leukemia, Acute, Childhood
Keywords: Relapsed Disease; MRD-positive CD19+ ALL; Natural History
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Retrospective chart review of children and adults with cancer enrolled on immunotherapy treatment protocols

SUMMARY:
Study Description:

This retrospective protocol focuses on characterizing clinical outcomes and toxicities following CAR T-cell therapy.

Objectives:

Primary

To evaluate the Response Free Survival (RFS) at 6 months following CD19 CAR stratified by prior blinatumomab vs no prior blinatumomab

To retrospectively evaluate outcomes following CAR T-cell therapy across children and young adults with B-ALL

Secondary

To evaluate the RFS at 12 months following CD19 CAR stratified by prior blinatumomab vs no prior blinatumomab and other immunotherapy.

To evaluate the incidence of CD19 negative versus CD19 positive relapse following CD19 CAR stratified by prior blinatumomab vs no prior blinatumomab.

To evaluate the Complete Response (CR) rate following CD19 CAR stratified by prior blinatumomab vs no prior blinatumomab.

To evaluate the Minimal Residual Disease (MRD) negative remission rate following CD19 CAR stratified by prior blinatumomab vs no prior blinatumomab.

Study Population and Source of Data: Subjects who were less than < 25 years of age at the time of diagnosis and received a CAR T-cell product for B-ALL.

DETAILED DESCRIPTION:
Study Description:

This retrospective protocol focuses on characterizing clinical outcomes and toxicities following CAR T-cell therapy.

Objectives:

Primary

To evaluate the Response Free Survival (RFS) at 6 months following CD19 CAR stratified by prior blinatumomab vs no prior blinatumomab

To retrospectively evaluate outcomes following CAR T-cell therapy across children and young adults with B-ALL

Secondary

To evaluate the RFS at 12 months following CD19 CAR stratified by prior blinatumomab vs no prior blinatumomab and other immunotherapy.

To evaluate the incidence of CD19 negative versus CD19 positive relapse following CD19 CAR stratified by prior blinatumomab vs no prior blinatumomab.

To evaluate the Complete Response (CR) rate following CD19 CAR stratified by prior blinatumomab vs no prior blinatumomab.

To evaluate the Minimal Residual Disease (MRD) negative remission rate following CD19 CAR stratified by prior blinatumomab vs no prior blinatumomab.

Study Population and Source of Data: Subjects who were less than < 25 years of age at the time of diagnosis and received a CAR T-cell product for B-ALL.

ELIGIBILITY:
* Subjects will not be recruited for this study; however, up to 210 subjects records will be selected from treatment protocols who received CAR therapy for B-ALL. Subject who opted out of the future use of his/her data will be excluded. The subjects enrolled to a CAR T cell therapy treatment protocol within the Pediatric Oncology Branch unless, are < 25 years of age at the time of diagnosis and must have received prior a CAR T-cell product.

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects who were < = 25 years of age at the time of diagnosis and received a CAR T-cell product for B-ALL. This protocol will be amended to incorporate new research objectives and new data as necessary
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
Outcome evaluation | 12 months
  To retrospectively evaluate outcomes following CAR T-cell therapy across children and young adults with B-ALL
Response free survival | 6 months
  To evaluate the RFS at 6 months following CD19 CAR stratified by prior blinatumomab vs no prior blinatumomab.

SECONDARY OUTCOMES:
Minimal Residual Disease detection | 12 months
  To evaluate the MRD negative remission rate following CD19 CAR stratified by prior blinatumomab vs no prior blinatumomab
Response free survival | 12 months
  To evaluate the RFS at 12 months following CD19 CAR stratified by prior blinatumomab vs no prior blinatumomab
Relapse Rate | 12 months
  To evaluate the incidence of CD19 negative versus CD19 positive relapse following CD19 CAR stratified by prior blinatumomab vs no prior blinatumomab
Complete Remission Rate | 12 months
  To evaluate the CR rate following CD19 CAR stratified by prior blinatumomab vs no prior blinatumomab

CONTACTS AND LOCATIONS:
Overall Officials: Nirali N Shah, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.